CLINICAL TRIAL: NCT01022749
Title: Prospective, Multicentre, Open-label Study Evaluating the Immunogenicity and Safety of Influenza Vaccine in Patients With Inflammatory Bowel Disease (IBD) Receiving or Not Immunosuppressive Therapy
Brief Title: Efficacy Safety Study of Flu Vaccine in Immunodepression Patients
Acronym: MICIVAX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Paris 5 - Rene Descartes (Other); Pierre and Marie Curie University (Other); Institut Pasteur (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P 070165
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: inflammatory bowel disease (IBD); immunosuppressed or non-immunosuppressed; influenza vaccine; antibody titers; seroprotective titers; vaccine-associated adverse events
MeSH Terms: conditions — Inflammatory Bowel Diseases; Influenza, Human | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 (Experimental): patients with IBD receiving immunosuppressants (TNF blockers excluded) (n=100)
  Interventions: Drug: Vaccine
- 3 (Experimental): patients with IBD receiving immunosuppressants including TNF blockers (n=100)
  Interventions: Drug: Vaccine
- 1 (Experimental): patients with IBD not receiving immunosuppressant (n=100)
  Interventions: Drug: Vaccine
- 4 (Active Comparator): patients with IBD receiving immunosuppressants including TNF blockers (n=20)
  Interventions: Biological: Vaccine anti-H1N1

INTERVENTIONS:
Drug: Vaccine — MUTAGRIP (2009-2010 winter) VAXIGRIP (2010-2011 winter)
  Arms: 1; 2; 3
Biological: Vaccine anti-H1N1 — patients who received the vaccine anti-H1N1
  Arms: 4

SUMMARY:
The primary purpose of the study is to compare the efficacy and safety of influenza vaccine in patients with inflammatory bowel disease (IBD) receiving immunosuppressive therapy with patients not receiving immunosuppressants .

The main objective of the study is to evaluate the humoral immunogenicity of influenza vaccination in patients with IBD

DETAILED DESCRIPTION:
Annual vaccination against influenza is recommended for those at high risk of complications, particularly among patients with immunodeficiency including those resulting from immunosuppressive treatments administered for a chronic inflammatory bowel disease (IBD). However, published data showing that influenza vaccination coverage is low in this population (<30%) due to lack of data on the effectiveness of vaccination in these patients and the theoretical risk of negative impact on the evolution of IBD.

To improve influenza vaccination coverage of the population treated by immunosuppressants for a chronic IBD, it is essential to have data on the effectiveness of vaccination in these populations.

The research aims to evaluate the immunogenicity of influenza vaccination in patients followed for a chronic IBD.

Factors in choice of study population were as follows:

1. IBD is a common disease. Among the inflammatory diseases treated with immunosuppressants and reaching patients under 65 years, IBD are among the most frequent. They result from an abnormal immune response to gut flora and their management often requires the prescription of immunosuppressive drugs (azathioprine, methotrexate, in particular) and more recently TNF-blockers;
2. the existence of vaccine recommendations published recently for specific patients on immunosuppressive therapy at greatest risk of complications related to influenza;
3. the fact that vaccinations have not been implicated in the pathogenesis of the disease;
4. data showing that vaccination recommendations are poorly followed in this population. A recently published work found vaccination coverage against influenza of only 28% in a cohort of 169 patients treated for IBD;

The methodology chosen is a phase III, prospective, open, vaccine trial. The primary endpoint is the humoral immunogenicity induced by the vaccine.

The study is scheduled on 2 successive years to assess the value of annual vaccination repeated in this population treated with immunosuppressants.

There is a benefit for patients to participate in this study because they are all vaccinated against influenza and will benefit from a clinical and laboratory monitoring in this study. Moreover, these patients are taken to be vaccinated in the event of a pandemic influenza

ELIGIBILITY:
Inclusion criteria :

* informed consent signed
* Age between 18 to 64
* Patient suffering from chronic inflammatory bowel disease (Crohn's disease, ulcerative colitis, or indeterminate colitis)
* For patients receiving at least one immunosuppressive or anti-TNF therapy: treatment introduced for at least 3 months
* Patient willing to participate in the study throughout its duration and acceptance procedures related to the study (blood samples, self questionnaires, nasal swab and telephone follow-up)

Exclusion criteria :

* Patient treated by corticosteroid alone without immunosuppressive or anti-TNF
* For women, being pregnant or positive pregnancy test
* Known allergy to any component of the study vaccine or a history of hypersensitivity reaction to influenza vaccination
* Fever (at least 37.5°C measured orally) or acute infection in the week prior to vaccination
* Received influenza vaccination in the 6 months preceding enrollment
* Known history of progressive neuropathy or Guillain-Barre
* Known infection with HIV and/or HBV (Ag-HBs positive) and/or HCV
* Other causes of severe immune deficiency
* Cellular therapy, immunoglobulin infusions, of blood products or monoclonal antibodies (except anti-TNF) in the 3 months prior to vaccination
* Patient deprived of freedom by an administrative or court order
* Patient non affiliated to a health social security system

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | 3-4 weeks after vaccination
  Seroconversion rate in the overall population, defined as the geometric mean titers ratio post / pre-vaccination for each of the three vaccine strains

SECONDARY OUTCOMES:
Seroconversion factor | 3 weeks and 6 months after vaccination
  The seroconversion factor obtained for each of the three vaccine strains will be compared between each of the three groups (patients not receiving treatment, patients receiving immunosuppressants and patients receiving immunosuppressants including TNF) defined as the geometric mean titers ratio post / pre-vaccination for each of the three vaccine strains
Seroprotection rate against the three vaccine strains | 3 or 4 weeks after of vaccination
  The seroprotection rate (defined as the proportion of subjects attaining an anti-hemagglutinin titer ≥1:40) obtained 3-4 weeks after flu vaccination, against the three vaccine strains
Seroprotection rate in the general population | 3 weeks and 6 months after vaccination
  The seroprotection rate in the general population and according to the three groups of patients
Seroconversion rate, geometric mean titers ratio before and after vaccination by haemagglutination inhibition assay | after 3 weeks of vaccination
  The seroconversion rate, geometric mean titers ratio before and after vaccination by haemagglutination inhibition (HI) assay before and after vaccination
Comparison of seroprotection rates for each of the three vaccine strains obtained in each of three groups | 3 weeks and 6 months of vaccination
  Comparison of seroprotection rates for each of the three vaccine strains obtained in each of three groups (patients not receiving treatment, patients receiving immunosuppressants and patients, receiving immunosuppressants including TNF)
Comparison of seroconversion factors obtained after 1 or 2 vaccinations in each of three groups of inflammatory bowel disease (IBD) and in the entire population | After 3 weeks of vaccination
Number of influenza episodes and confirmed flu during each influenza peak season | 6 months after vaccination
Occurrence of medical visits, emergency room visits, hospital admissions and deaths throughout the course of the study | 18 months after vaccination
Occurrence and intensity of local and general adverse events within 5 days after vaccine administration | 5 days after vaccination
Search of the determining factors to the influenza vaccine response | 18 months after vaccination
  Search of the determining factors to the influenza vaccine response: sex, age, previous vaccination against influenza, chronic smoking, the presence of other comorbidities (diabetes, renal failure, cirrhosis, ..), the nature of the IBD, the nature of the treatment of IBD and their duration, the number of immunosuppressive treatments associated and Disease Activity Index score of IBD at the vaccination time
Sub-immunological study | 6 months after vaccination
  Sub-immunological study each year of the study, the first and the second year (n=60, 20 patients per group): To determine if the LT-CD4 induction at J21-28 is correlated with the antibody anti-vaccines concentration measured within 6 months. To determine if the basal concentrations of anti-flu LT-CD4 at J21-J28 is correlated with the antibody anti-vaccines concentrations measured within 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Odile LAUNAY, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CIC Vaccinologie Hopital Cochin, Paris, France

REFERENCES:
- [Result] Loison E, Poirier-Beaudouin B, Seffer V, Paoletti A, Abitbol V, Tartour E, Launay O, Gougeon ML. Suppression by thimerosal of ex-vivo CD4+ T cell response to influenza vaccine and induction of apoptosis in primary memory T cells. PLoS One. 2014 Apr 1;9(4):e92705. doi: 10.1371/journal.pone.0092705. eCollection 2014. PMID 24690681
- [Derived] Launay O, Abitbol V, Krivine A, Slama LB, Bourreille A, Dupas JL, Hebuterne X, Savoye G, Deplanque D, Bouhnik Y, Pelletier AL, Galtier F, Laharie D, Nachury M, Zerbib F, Allez M, Bommelaer G, Duclos B, Lucht F, Gougeon ML, Tartour E, Rozenberg F, Hanslik T, Beaugerie L, Carrat F; MICIVAX Study Group. Immunogenicity and Safety of Influenza Vaccine in Inflammatory Bowel Disease Patients Treated or not with Immunomodulators and/or Biologics: A Two-year Prospective Study. J Crohns Colitis. 2015 Dec;9(12):1096-107. doi: 10.1093/ecco-jcc/jjv152. Epub 2015 Sep 7. PMID 26351392